CLINICAL TRIAL: NCT05949710
Title: Explore the Relationship Between Heart Rate Variability, Body Mass Index, Inflammation, and Insulin Resistance: From a Population-based Survey to Multi-arms of Aerobic Exercise Intervention.
Brief Title: Explore the Relationship Between Heart Rate Variability, Body Mass Index, Inflammation, and Insulin Resistance.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Tainan Junior College of Nursing (Other)
Responsible Party: Principal Investigator, Yu-Hsuan Chang, Assistant professor, National Tainan Junior College of Nursing
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NTJCN
Record Dates: First submitted 2023-06-28; First posted 2023-07-18 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Obesity; Insulin Resistance; Overweight
Keywords: heart rate variability; exercise; inflammation; insulin resistance
MeSH Terms: conditions — Obesity; Insulin Resistance; Overweight; Motor Activity; Inflammation | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Particiapnts will be divided into two groups: normal weight group and overweight/obese group.
Who Masked: Outcomes Assessor
Masking Description: The data analyzer (PI) will be blinded but the participants and intervener will not be.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aerobic exercise(AE), normal weight (Experimental): 3 times a week, normal weight
  Interventions: Behavioral: aerobic exercise(AE)
- aerobic exercise(AE) , overweight/obese (Experimental): 3 times a week, overweight/obese
  Interventions: Behavioral: aerobic exercise(AE)

INTERVENTIONS:
Behavioral: aerobic exercise(AE) — The participants will receive AE three times per week.

SUMMARY:
The findings will serve as a reference for clinical professionals to promote exercise among the general population for improving HRV.

DETAILED DESCRIPTION:
Background: Heart rate variability (HRV) measurement is widely used to assess the function of cardiac autonomic modulation. Aerobic exercise (AE) has been proven to improve HRV. However, because HRV is highly associated with visceral fat, inflammatory status, and insulin resistance, whether baseline body inflammation status can explain the heterogeneous response to AE remains unknown.

Purposes: We will compare the effects of AE training in improving HRV, inflammatory markers, and insulin resistance between community residents with normal weight and overweight/obesity.

Methods: A quasi-experimental study with purposive sampling will be used to recruit community residents aged 40-64 years with inactive habits in southern Taiwan. The minimum targeted sample size is 43 participants. The participants will be grouped into normal weight and overweight/obese groups. All participants will receive AE training with at least moderate intensity three times per week. HRV parameters, blood samples, and visceral fat will be evaluated. The blood samples will be evaluated for C-reactive protein and markers of insulin resistance (fasting glucose, insulin). All participants will be evaluated at baseline (T0) and after a 16-week intervention (T1). In addition to these time points, HRV will be measured during every exercise session for participants in exercise groups. Generalized estimating equations will be used to determine whether baseline BMI is the key factor influencing the effects of AE.

Relevance to clinical practice: The findings will serve as a reference for clinical professionals to promote exercise among the general population for improving HRV.

ELIGIBILITY:
Inclusion Criteria:

* are aged between 40 and 64 years.
* had inactive habit (<3 days of physical activity per week and <30 minutes per session).
* can communicate in Mandarin or Taiwanese.

Exclusion Criteria:

* underlying conditions, such as stroke, acute coronary artery diseases, handicap, pregnancy, and unstable hypertension, that may present risks for exercise training.
* smoking or alcohol abuse.
* currently being on a diet, and (d) lifestyles that may affect HRV and inflammatory biomarkers (e.g., shift work or habit of staying up late).

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Compared to men, women tends to engage in community activities in Taiwan.
Enrollment: 51 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | two times and each session of exercise (change from baseline to the end of 16-week)
  will use heart rate variability analyzer
insulin resistance | two times (change from baseline to the end of 16-week)
  μIU/mL
Visceral fat | two times (change from baseline to the end of 16-week)
  will use body composition analyzer
fasting glucose | two times (change from baseline to the end of 16-week)
  mg/dL
C-reactive protein | two times (change from baseline to the end of 16-week)
  mg/L
Waist-to-hip ratio | two times (change from baseline to the end of 16-week)
  Waist-to-hip ratio
Waist-to-height ratio | two times (change from baseline to the end of 16-week)
  Waist-to-height ratio
body weight | two times (change from baseline to the end of 16-week)
  weight in Kilogram
BMI | two times (change from baseline to the end of 16-week)
  weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsuan Chang, phD, Principal Investigator — National Tainan Junior College of Nursing
Locations (1):
- Yu-Hsuan Chang, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No
for research privacy.